CLINICAL TRIAL: NCT05573347
Title: Comparison of the Cellular Content of Bone Marrow Aspiration From the Posterior Superior Iliac Spine and Deep Humeral Harvest in Patients Undergoing Rotator Cuff Repair
Brief Title: Cellular Content of Bone Marrow Aspiration, Comparison
Acronym: BioCuff
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Andrews Research & Education Foundation (Other)
Collaborators: Florida (Other)
Responsible Party: Sponsor
Other Study IDs: RC Comp (BioCuff)
Record Dates: First submitted 2022-10-03; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Rotator Cuff Tear or Rupture, Not Specified as Traumatic
MeSH Terms: conditions — Rotator Cuff Injuries; Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone marrow aspirate from harvest
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bone marrow harvest from side-lying patient: This group will have bone marrow harvested from the PSIS extraction site while lying in the lateral decubitus position.
  Interventions: Procedure: Rotator Cuff Repair; Procedure: Bone Marrow Harvest
- Bone marrow harvest from patient lying prone: This group will have bone marrow harvested from the PSIS extraction site while lying in the prone position.
  Interventions: Procedure: Rotator Cuff Repair; Procedure: Bone Marrow Harvest

INTERVENTIONS:
Procedure: Rotator Cuff Repair — Surgical repair of one or more ligament(s) that form the rotator cuff shoulder complex (supraspinatus, infraspinatus, subscapularis, and teres minor)
Procedure: Bone Marrow Harvest — Procedure in which bone marrow cells are extracted, or harvested, from a given location in the body
  Other Names: Bone Marrow Aspiration

SUMMARY:
The goal of this observational clinical trial is to determine whether the posterior superior iliac spine of the hip or the humerus of the arm will produce larger amounts of bone marrow when harvested during surgery. Also, the secondary goal of this study is to determine the effects of the patient's position on the quantity of cells harvested from the hip, namely lying on back (prone) vs. lying on side (lateral decubitus). The main questions it aims to answer are:

* Will the hip or the arm have more bone marrow extracted?
* Does a patient lying in lateral decubitus position produce more bone marrow than lying in the prone position?

Participants that are to undergo rotator-cuff repair are eligible for this study. During the participant's repair, bone marrow will be extracted from the arm and from the hip. Half of the eligible participants will have bone marrow extracted from the hip while lying on their side, while the other half will have bone marrow extracted from the hip while lying on their back. Researchers will compare the results from both extraction sites on each patient, as well as compare results of the two patient position groups.

DETAILED DESCRIPTION:
This is a single site, comparative quantitative analysis study of the cellular characteristics of bone marrow aspirate from two extraction sites (PSIS and humerus) from patients undergoing standard-of-care arthroscopic rotator cuff repair surgery. 30 total patients will be recruited through the Andrews Institute physician practices. A recruitment flyer will be used to recruit participants. The flyer will be placed within physicians' offices and on social media platforms. Potential participants will be prescreened for inclusion and exclusion criteria through standard of care medical evaluations. Once a potential participant has agreed to be involved in the study, they will go through the described informed consent process. Patients meeting the inclusion criteria will have the study explained to them by one of the members of the research team, and they will be given an opportunity to participate if they are interested.

After the described screening and informed consent process have been completed, all participants will undergo standard-of-care arthroscopic rotator cuff repair surgery. During all surgeries, bone marrow will be aspirated from the PSIS and from the humerus. The first 15 participants will have bone marrow aspirated from the PSIS while in the prone position on the operating table. The final 15 participants will have bone marrow aspirated from the PSIS while in the lateral decubitus position on the operating table. Both cohorts will undergo humeral harvest intraoperatively in the lateral decubitus position. One mL of concentrated bone marrow aspirate (cBMA) from each harvest site from each surgery will be removed and sent to the AREF Regenerative Medicine Center (RMC) for analysis. The remaining cBMA will be used to augment the rotator cuff repair surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age
* Diagnosis of a rotator cuff tear requiring arthroscopic rotator cuff repair

Exclusion Criteria:

* Patients who require superior capsular reconstruction or revision rotator cuff repair
* Diabetes
* Immune Disorders
* Past medical history of a metastatic or other cancer which required chemotherapy/ radiation therapy
* Rheumatoid arthritis
* Is unable to comprehend the study documents or give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The focus demographic of this study is people within the ages of 18 and 80 that have been diagnoses with a rotator cuff tear and require reconstructive surgery.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2023-08-16 (Estimated); Study Completion 2023-08-16 (Estimated)

PRIMARY OUTCOMES:
Hemocytometer (Sysmex) | Upon day of surgical procedure (once per participant)
  Machine that separates blood cells into categories, including red blood cell (RBC), white blood cell (WBC), monocyte, platelet, and hematopoietic progenitor cell (HPC) groups to assess concentration

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Hackel, MD, Principal Investigator — Orthopedic Surgeon
Locations (1):
- Andrews Research and Education Foundation, Gulf Breeze, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akpancar S, Tatar O, Turgut H, Akyildiz F, Ekinci S. The Current Perspectives of Stem Cell Therapy in Orthopedic Surgery. Arch Trauma Res. 2016 Aug 16;5(4):e37976. doi: 10.5812/atr.37976. eCollection 2016 Dec. PMID 28144608
- [Background] Marycz K, Mierzejewska K, Smieszek A, Suszynska E, Malicka I, Kucia M, Ratajczak MZ. Endurance Exercise Mobilizes Developmentally Early Stem Cells into Peripheral Blood and Increases Their Number in Bone Marrow: Implications for Tissue Regeneration. Stem Cells Int. 2016;2016:5756901. doi: 10.1155/2016/5756901. Epub 2015 Nov 9. PMID 26664409
- [Background] Rochefort GY, Delorme B, Lopez A, Herault O, Bonnet P, Charbord P, Eder V, Domenech J. Multipotential mesenchymal stem cells are mobilized into peripheral blood by hypoxia. Stem Cells. 2006 Oct;24(10):2202-8. doi: 10.1634/stemcells.2006-0164. Epub 2006 Jun 15. PMID 16778152
- [Background] Hauser RA, Orlofsky A. Regenerative injection therapy with whole bone marrow aspirate for degenerative joint disease: a case series. Clin Med Insights Arthritis Musculoskelet Disord. 2013 Sep 4;6:65-72. doi: 10.4137/CMAMD.S10951. eCollection 2013. PMID 24046512
- [Background] Hernigou P, Flouzat Lachaniette CH, Delambre J, Zilber S, Duffiet P, Chevallier N, Rouard H. Biologic augmentation of rotator cuff repair with mesenchymal stem cells during arthroscopy improves healing and prevents further tears: a case-controlled study. Int Orthop. 2014 Sep;38(9):1811-8. doi: 10.1007/s00264-014-2391-1. Epub 2014 Jun 7. PMID 24913770
- [Background] Hernigou P, Poignard A, Zilber S, Rouard H. Cell therapy of hip osteonecrosis with autologous bone marrow grafting. Indian J Orthop. 2009 Jan;43(1):40-5. doi: 10.4103/0019-5413.45322. PMID 19753178
- [Background] Hernigou P, Poignard A, Beaujean F, Rouard H. Percutaneous autologous bone-marrow grafting for nonunions. Influence of the number and concentration of progenitor cells. J Bone Joint Surg Am. 2005 Jul;87(7):1430-7. doi: 10.2106/JBJS.D.02215. PMID 15995108
- [Background] Saw KY, Anz A, Siew-Yoke Jee C, Merican S, Ching-Soong Ng R, Roohi SA, Ragavanaidu K. Articular cartilage regeneration with autologous peripheral blood stem cells versus hyaluronic acid: a randomized controlled trial. Arthroscopy. 2013 Apr;29(4):684-94. doi: 10.1016/j.arthro.2012.12.008. Epub 2013 Feb 4. PMID 23380230
- [Background] Vangsness CT Jr, Sternberg H, Harris L. Umbilical Cord Tissue Offers the Greatest Number of Harvestable Mesenchymal Stem Cells for Research and Clinical Application: A Literature Review of Different Harvest Sites. Arthroscopy. 2015 Sep;31(9):1836-43. doi: 10.1016/j.arthro.2015.03.014. PMID 26354202
- [Background] Kitoh H, Kitakoji T, Tsuchiya H, Katoh M, Ishiguro N. Transplantation of culture expanded bone marrow cells and platelet rich plasma in distraction osteogenesis of the long bones. Bone. 2007 Feb;40(2):522-8. doi: 10.1016/j.bone.2006.09.019. Epub 2006 Oct 27. PMID 17070744
- [Background] Ellera Gomes JL, da Silva RC, Silla LM, Abreu MR, Pellanda R. Conventional rotator cuff repair complemented by the aid of mononuclear autologous stem cells. Knee Surg Sports Traumatol Arthrosc. 2012 Feb;20(2):373-7. doi: 10.1007/s00167-011-1607-9. Epub 2011 Jul 20. PMID 21773831
- [Background] Hyer CF, Berlet GC, Bussewitz BW, Hankins T, Ziegler HL, Philbin TM. Quantitative assessment of the yield of osteoblastic connective tissue progenitors in bone marrow aspirate from the iliac crest, tibia, and calcaneus. J Bone Joint Surg Am. 2013 Jul 17;95(14):1312-6. doi: 10.2106/JBJS.L.01529. PMID 23864180
- [Background] Pierini M, Di Bella C, Dozza B, Frisoni T, Martella E, Bellotti C, Remondini D, Lucarelli E, Giannini S, Donati D. The posterior iliac crest outperforms the anterior iliac crest when obtaining mesenchymal stem cells from bone marrow. J Bone Joint Surg Am. 2013 Jun 19;95(12):1101-7. doi: 10.2106/JBJS.L.00429. PMID 23783207
- [Background] Beitzel K, McCarthy MB, Cote MP, Durant TJ, Chowaniec DM, Solovyova O, Russell RP, Arciero RA, Mazzocca AD. Comparison of mesenchymal stem cells (osteoprogenitors) harvested from proximal humerus and distal femur during arthroscopic surgery. Arthroscopy. 2013 Feb;29(2):301-8. doi: 10.1016/j.arthro.2012.08.021. Epub 2013 Jan 3. PMID 23290182
- [Background] Marx RE, Tursun R. A qualitative and quantitative analysis of autologous human multipotent adult stem cells derived from three anatomic areas by marrow aspiration: tibia, anterior ilium, and posterior ilium. Int J Oral Maxillofac Implants. 2013 Sep-Oct;28(5):e290-4. doi: 10.11607/jomi.te10. PMID 24066346
- [Background] Vasiliadis AV, Galanis N. Human bone marrow-derived mesenchymal stem cells from different bone sources: a panorama. Stem Cell Investig. 2020 Aug 10;7:15. doi: 10.21037/sci-2020-013. eCollection 2020. PMID 32964008
- [Background] Anz A, Sherman B. Concentrated Bone Marrow Aspirate Is More Cellular and Proliferative When Harvested From the Posterior Superior Iliac Spine Than the Proximal Humerus. Arthroscopy. 2022 Apr;38(4):1110-1114. doi: 10.1016/j.arthro.2021.10.011. Epub 2021 Oct 26. PMID 34715280
- [Background] Oliver K, Awan T, Bayes M. Single- Versus Multiple-Site Harvesting Techniques for Bone Marrow Concentrate: Evaluation of Aspirate Quality and Pain. Orthop J Sports Med. 2017 Aug 29;5(8):2325967117724398. doi: 10.1177/2325967117724398. eCollection 2017 Aug. PMID 28890905

DOCUMENTS (2):
  • Study Protocol (2022-08-12): https://cdn.clinicaltrials.gov/large-docs/47/NCT05573347/Prot_000.pdf
  • Informed Consent Form (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/47/NCT05573347/ICF_001.pdf